CLINICAL TRIAL: NCT02174198
Title: The Esthetic Effect of Bio-OSS Collagen® on the Mid-facial Gingival Dimensions When Placed Into Gaps Between 3i® Implants Placed Into Fresh Extraction Sockets and the Labial Plate of Bone
Brief Title: Bone Remodeling After Immediate Implant Placement With and Without Bone Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Principal Investigator, Nurit Bittner Fogel, Assistant Professor of Dental Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAM4053
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Results first posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-05

CONDITIONS: Tooth Loss
Keywords: Immediate implant; bone graft; immediate restoration
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BioOss Collagen (Experimental): Intervention: BioOss Collagen at the time of implant placement
  Interventions: Device: BioOss Collagen at the time of implant placement
- No Bone Graft (No Intervention): No placement of BioOss at the time of implant placement

INTERVENTIONS:
Device: BioOss Collagen at the time of implant placement — Experimental: placement of BioOss Collagen No intervention: no BioOss Collagen
  Other Names: BioOss Collagen, Geistlich Pharma Inc.
  Arms: BioOss Collagen

SUMMARY:
This study compares two ways of placing a dental implant on the day of tooth extraction. One method will place a additional bone graft (derived from bovine bone) and the other group will not have the graft placed. Both groups will be restored at the same time with an immediate crown.

The investigators will be researching and comparing the changes in gum level that occur after each surgical method, as well as changes in jaw width where the implant is placed.

The investigators will enroll 16 patients per group. The patients will be followed for 3, 6, and 12 months post-immediate implant placement to observe healing.

DETAILED DESCRIPTION:
The purpose of the current study is to evaluate the soft tissue dimensional changes after extraction of teeth in the esthetic zone, when combined with the placement of implants into these fresh extraction sockets. In addition, the effect of placing a graft material, such as Bio-Oss Collagen® into the gap between implant and the labial plate of bone will be evaluated after an immediately loaded provisional restoration is placed. 32 subjects will have an immediate dental implant placed in the maxillary anterior region (#4-12) after extraction of a hopeless tooth. 16 subjects will be randomly selected to receive Bio-Oss Collagen® (Test group) and 16 subjects will have no graft (Control group) in the gap between the implant and the labial plate of bone. Hopeless maxillary anterior teeth will be extracted and implants will be placed in a flapless procedure. Implants will be immediately loaded with provisional restorations once determined that the implant is stable. Changes in vertical height and horizontal dimensional changes of the free gingival margins will be evaluated at 3, 6, and 12 months post-immediate implant placement.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have read, understood and signed an informed consent form.
2. Subjects must be willing and able to follow study procedures and instructions.
3. Subjects must have labial plate of bone present after extraction no more than 4 mm from the free gingival margin.
4. Subjects must require one maxillary anterior implant.
5. Subjects must be older than 18 years

Exclusion Criteria:

1. Subjects having participated within the last six months in other clinical studies.
2. Subjects who have failed to maintain good plaque control.
3. Subjects with any systemic condition like uncontrolled diabetes mellitus, cancer, human immunodeficiency virus (HIV), disorders that compromise wound healing, chronic high dose steroid therapy, bone metabolic diseases, radiation or other immuno-suppressive therapy which would preclude periodontal surgery.
4. Subjects with the presence of acute infectious lesions in the areas intended for surgery.
5. History within the last 6 months of weekly or more frequent use of smokeless chewing tobacco, pipe or cigar smoking and cigarette smoking (greater than 10 cigarettes per day).
6. Female subjects who are pregnant or lactating, or who intend to become pregnant during the study period following entrance into the study.
7. Subjects on Bisphosphonate Therapy with C-terminal telopeptide (CTX) values <100
8. Subjects requiring antibiotic prophylaxis for subacute bacterial endocarditis (SBE) or late prosthetic joint infection. Patients who cannot undergo standard oral surgery procedure for any reason.
9. Subjects that have adjacent teeth next to tooth slated for extraction and immediate placement showing periodontal disease, endodontic and/or caries pathology will be excluded.
10. Subjects having unfavorable occlusal schemes for immediate loading, parafunctional habits and inadequate posterior support to properly protect the anterior teeth during function.
11. Implant site will not be next to an adjacent implant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nurit Bittner Fogel, DDS, Principal Investigator — Columbia University
Locations (1):
- Columbia University, College of Dental Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BioOss Collagen | No Bone Graft
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BioOss Collagen | No Bone Graft | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (4.2) | 52.3 (3.3) | 52.3 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 12 | 8 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 8 | 12
Number of Smokers [Count of Participants; unit: Participants] | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Bucco-Lingual Change at 3mm
Description: The horizontal dimensional change from a digital superimposition at 3mm apical to the baseline free gingival margin position was measured.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | BioOss Collagen | No Bone Graft
Number analyzed (Participants) | 16 | 16
mm | -0.84 (0.64) | -1.01 (0.45)

2. Primary Outcome: Mean Bucco-Lingual Change at 4mm
Description: The horizontal dimensional change from a digital superimposition at 4mm apical to the baseline free gingival margin position was measured.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | BioOss Collagen | No Bone Graft
Number analyzed (Participants) | 16 | 16
mm | -0.64 (0.62) | -0.80 (0.33)

3. Secondary Outcome: Change in Vertical Dimension of Buccal Soft Tissue (Distal Papilla)
Description: The mean change was calculated from a tooth-supported stent to the free gingival margin.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | BioOss Collagen | No Bone Graft
Number analyzed (Participants) | 16 | 16
mm | -0.4 (1.2) | -1.4 (1.1)

4. Secondary Outcome: Change in Vertical Dimension of Buccal Soft Tissue (Mid-buccal)
Description: The mean change was calculated from a tooth-supported stent to the free gingival margin.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | BioOss Collagen | No Bone Graft
Number analyzed (Participants) | 16 | 16
mm | -0.9 (1.2) | -1.3 (1.5)

5. Secondary Outcome: Change in Vertical Dimension of Buccal Soft Tissue (Mesial Papilla)
Description: The mean change was calculated from a tooth-supported stent to the free gingival margin.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | BioOss Collagen | No Bone Graft
Number analyzed (Participants) | 16 | 16
mm | -0.6 (1.2) | -0.9 (1.4)

6. Secondary Outcome: Periodontal Probing Depth
Description: The periodontal probing depth will be measured in mm.
Time Frame: 12 months
Population: Data for this outcome measure was not collected and analyzed since all the patients on the study were periodontally healthy and showed no signs of soft tissue inflammation.
Arm/Group | BioOss Collagen | No Bone Graft
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Thickness of Keratinized Tissue at 3mm
Description: Tissue thickness was measured at 3mm from the free gingival margin (FGM) using a 15-endodontic file and a rubber stopper.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | BioOss Collagen | No Bone Graft
Number analyzed (Participants) | 16 | 16
mm | 1.7 (0.6) | 1.7 (0.7)

8. Secondary Outcome: Thickness of Keratinized Tissue at 4mm
Description: Tissue thickness was measured at 4mm from the free gingival margin (FGM) using a 15-endodontic file and a rubber stopper.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | BioOss Collagen | No Bone Graft
Number analyzed (Participants) | 16 | 16
mm | 1.4 (0.4) | 1.6 (0.8)

9. Secondary Outcome: Thickness of Keratinized Tissue at 8mm
Description: Tissue thickness was measured at 8mm from the free gingival margin (FGM) using a 15-endodontic file and a rubber stopper.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | BioOss Collagen | No Bone Graft
Number analyzed (Participants) | 16 | 16
mm | 1.5 (0.5) | 1.8 (0.8)

ADVERSE EVENTS:
Time Frame: From baseline to 12 months.
Arm/Group | BioOss Collagen | No Bone Graft
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

LIMITATIONS AND CAVEATS:
The sample size for this study is limited, as well as the overall follow up of the patients. Further, studies with longer follow up times may be recommended to evaluate long term behavior of the tissues with immediately placed implants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT02174198/Prot_SAP_000.pdf